CLINICAL TRIAL: NCT07102108
Title: A Prospective Observational Study on the Effects of Anesthesia Techniques on Tissue Oxygenation and Postoperative Recovery in Lower Abdominal Surgery
Brief Title: Effects of Anesthesia Techniques on Tissue Oxygenation and Recovery in Lower Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Ars Gor Dr Edip Gules, Research Assistant-Anestesthesiology and Reanimation, Trakya University
Other Study IDs: TUTF-GOBAEK 2023-25; TUTF-GOBAEK 2023-25 (Other: Trakya University/Faculty of Medicine Ethics Committee)
Record Dates: First submitted 2025-07-03; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Lower Abdominal Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- General Anesthesia: Patient receiving general anesthesia only for lower abdominal surgery
- General+Epidural Anesthesia: Patient receiving combined general and epidural anesthesia for lower abdominal surgery
- Spinal: Patient receiving spinal anesthesia only for lower abdominal surgery
- Epidural Anesthesia: Patient receiving epidural anesthesia only for lower abdominal surgery

SUMMARY:
This is a prospective observational study designed to evaluate the effects of different anesthesia techniques on tissue oxygenation and postoperative recovery in patients undergoing lower abdominal surgery. A total of 180 patients will be enrolled and evenly allocated into four groups based on the anesthesia method used: general anesthesia, spinal anesthesia, epidural anesthesia, and combined general plus epidural anesthesia.

Near-infrared spectroscopy (NIRS) will be utilised to monitor tissue oxygenation at the thenar and plantar regions during the perioperative period. Vital signs, VAS scores(min 0-max 10 points), Quality of Recovery-40 (QoR-40) scores(min 40-max 200 points), and additional postoperative recovery parameters- including length of stay in the post-anesthesia care unit and hospital, surgical site infection, wound revision, and mortality- will be recorded and compared across the groups.

The primary hypothesis is that regional anesthesia techniques enchance tissue oxygenation and are associated with improved postoperative recovery outcomes compared to general anesthesia alone. The study was approved by the local ethics committee and will be conducted at a single tertiary-care center.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years
* Scheduled for elective lower abdominal surgery
* Eligible for general, spinal, epidural or combined anesthesia techniques
* Provided writen informed consent
* ASA physical status 1-3

Exclusion Criteria:

* Refusal to participate
* Emergency surgery
* Severe cardiovascular or respiratory instability
* Pre-existing severe cognitive impairment of communication barrier
* Peripheral vascular disease affecting NIRS readind
* Local infection or anatomical anomaly preventing regional anesthesia

Ages: 18 Days to 80 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adult patients aged 18-80 undergoing elective lower abdominal surgeries under one of four anesthesia techniques (general, spinal, epidural, or combined general+epidural) at a single tertiary hospital. Patients with peripheral vascular disease, severe cardiopulmonary instability, or cognitive/communication limitations were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Tissue Oxygenation Levels Measured by NIRS | From baseline(pre-op) to end of surgery
  Continuous measurement of tissue oxygenation at thenar and plantar sites using near-infrared spectroscopy during perioperative period

SECONDARY OUTCOMES:
Intraoperative Vital Signs | Intraoperative period
  Systolic blood pressure recorded during anesthesia
Intraoperative Vital Signs | Intraoperative period
  Diastolic blood pressure recorded during anesthesia
Intraoperative Vital Signs | Intraoperative period
  Heart rate recorded during anesthesia
Intraoperative Vital Signs | Intraoperative period
  Oxygenation saturation recorded during anesthesia
Visual Analog Scale(VAS) Pain Scores | Up to 24 hours after surgery
  VAS pain scores measured postoperatively at PACU and postoperative day 1. The scale ranges from 0 to 10, where 0 indicates no pain and 10 indicates the worst possible pain. Higher scores indicate worse outcomes.
Qor-40 Questionnaire Scores | postoperative day 1
  Quality of Recovery scores assessed using the Qor-40 questionnaire on postoperative day1. The total score ranges from 40 to 200, with higher scores indicating better recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Faculty of Medicine, Edirne, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No